CLINICAL TRIAL: NCT00710450
Title: The Effect of Montelukast In-vitro on Basophil Histamine and Leukotriene, IL-4 Adn IL-13 Release in Subjects With Allergic Rhinitis or Allergic Asthma
Brief Title: Effect of Montelukast on Basophils, In-vitro
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Creighton University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Townley Merck
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Asthma; Allergic Rhinitis
Keywords: IL13; leukotriene; histamine; IL4; Must be allergic asthma or allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Supernatents from stimulation assays will be kept for batch assay.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Allergic Asthma
- 2: Allergic Rhinitis

SUMMARY:
Subjects with either allergic asthma or allergic rhinitis will be recruited to obtain blood. This blood will be used to be stimulated with to whatever the patient allergic. In the laboratory, this stimulated blood will be measured for histamine, leukotrienes, IL-13 and IL-3. These are chemicals responsible for allergy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthma or allergic rhinitis
* age 12+

Exclusion Criteria:

* smokers

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Allergic rhinitis or allergic asthma, age 13+
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Histamine Release | during the assay portion.

SECONDARY OUTCOMES:
Cytokine release. IL-13, IL-4 and leukotriene | assay portion

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States